CLINICAL TRIAL: NCT05072340
Title: Evaluation of Resilience Skills Enhancement (RISE) Training Among University Students: A Sequential Mixed Methods Study
Brief Title: Evaluation of Resilience Skills Enhancement (RISE) Training Among University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Lau Ying, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TEG AY2021/22
Record Dates: First submitted 2021-08-11; First posted 2021-10-08 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Resilience, Psychological; Adaptation, Psychological
Keywords: Resilience training; Blended learning; Randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The allocation was done based on the participants' sequence of enrolment, and another research assistant opened the opaque envelopes and allocated participants to either the blended or self-guided RISE group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RISE (Blended learning) (Experimental): Students will undergo a training that comprises of six sessions: (1) introducing resilience, (2) coping strategies, (3) creating positivity, (4) shifting mindsets, (5) building social competency and (6) preparing for the future.
  RISE training will be hosted via the NUS' online learning platform, LumiNUS and virtual face-to-face platform, Zoom. Each session will take approximately one to two hours per week. One session is made available each week to encourage completion before moving onto the next session. Students will be provided with materials in the form of interactive videos. Virtual face-to-face sessions, online forum, quizzes and homework will be additionally available to students.
  Interventions: Behavioral: Resilience Skills Enhancement (RISE)
- RISE (Asynchronous learning) (Active Comparator): Students will also undergo a six-session training comprising of: (1) introducing resilience, (2) coping strategies, (3) creating positivity, (4) shifting mindsets, (5) building social competency and (6) preparing for the future.
  RISE training will be hosted via the NUS' online learning platform, LumiNUS. One session is made available each week to encourage completion before moving onto the next session. Participants will be reminded via emails and short message service (SMS) to complete the intervention. Students will be provided with materials in the form of interactive videos in LumiNUS.
  Interventions: Behavioral: Resilience Skills Enhancement (RISE)

INTERVENTIONS:
Behavioral: Resilience Skills Enhancement (RISE) — The RISE training was developed according to theory, empirical evidence and contextual information. The contents, components, pedagogy, and technical elements of RISE is established based on the resilience theory (Szanton & Gill, 2010) systematic review and meta-analysis, meta-synthesis, and qualitative study (Ang et al., 2021). Ethical and quality standards was assessed using the Health on the Net code of conduct and the Health-Related Website Evaluation Form respectively. The overall rating of the designed RISE is more than 75% of the total possible points to ensure quality of website by three research team members.

SUMMARY:
Background University students experience high levels of stress and this may negatively impact their mental health, coping and academic outcomes. Building resilience has been described as an ability to maintain mental well-being.

Aims This study aims to (1) assess the feasibility of the Resilience Skills Enhancement (RISE) program, (2) evaluate the effects of RISE on undergraduate students' resilience, coping, emotion regulation, positive emotions and stress and (3) explore students' perception of RISE.

Methods This study will be operationalized in three phases.

Phase 1 - Feasibility A single-arm pre-post study will be used. 10 students will be recruited to explore their acceptability, perception, and suggestions for improving RISE. RISE comprises of six weekly sessions delivered via LumiNUS and Zoom. The Wilcoxon signed rank test will be used to analyse the data.

Phase 2 - Randomized controlled trial A prospective, double blind randomized controlled trial and repeated post-tests will be used. A total of 122 students will be recruited from LumiNUS and social media platforms. Participants will receive a series of six, weekly online sessions in both groups. The primary outcome is resilience. The secondary outcomes include, coping, emotion relation, positive emotions, stress. Multivariate analysis of variance with repeated measures will be used to compare the mean difference of scores in the three time points through Wilks's lambda test. The data will be analysed according to the intention-to-treat principle.

Phase 3 - Process evaluation A qualitative study using an individual, semi-structured interviews will be used to explore students' perception of RISE. Approximately 20 students will be recruited, and the final sample size will be determined based on data saturation. Thematic analyses will be used to analyse the data.

Potential contributions This study will contribute by evaluating evidence-based user-friendly RISE that may be effective for enhancing university students' resilience.

ELIGIBILITY:
Inclusion Criteria:

1. Full undergraduate in NUS
2. Above 18 years old
3. Comprehend English language
4. Have access to an electronic device (laptop, smartphone or tablet)

Exclusion Criteria:

1. No self-reported history of mental health disorders
2. Did not participate in any other form of resilience training

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Resilience | Baseline
  Resilience will be measured using the 25-item Connor-Davidson Resilience Scale (CD-RISC, Connor & Davidson 2003). Items are rated on a 5-point Likert scale ranging from 0 (not true at all) to 4 (true nearly all the time), with higher scores indicating higher resilience. The CD-RISC has good psychometric properties (Windle et al., 2011) and validated among Singapore students (Chue & Cheung, 2021).
Resilience | After training complete
  Resilience will be measured using the 25-item Connor-Davidson Resilience Scale (CD-RISC, Connor & Davidson 2003). Items are rated on a 5-point Likert scale ranging from 0 (not true at all) to 4 (true nearly all the time), with higher scores indicating higher resilience. The CD-RISC has good psychometric properties (Windle et al., 2011) and validated among Singapore students (Chue & Cheung, 2021).
Resilience | Three months after training completes
  Resilience will be measured using the 25-item Connor-Davidson Resilience Scale (CD-RISC, Connor & Davidson 2003). Items are rated on a 5-point Likert scale ranging from 0 (not true at all) to 4 (true nearly all the time), with higher scores indicating higher resilience. The CD-RISC has good psychometric properties (Windle et al., 2011) and validated among Singapore students (Chue & Cheung, 2021).

SECONDARY OUTCOMES:
Social support | Baseline
  Social support will be measured using the Multidimensional Scale of Perceived Social Support Scale (MSPSS, Zimet et al., 1988). Items are rated on a 7-point Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree), with higher scores indicating better social support. The MSPSS has good psychometric properties and used among students (Dambi et al., 2018).
Social support | After training completes
  Social support will be measured using the Multidimensional Scale of Perceived Social Support Scale (MSPSS, Zimet et al., 1988). Items are rated on a 7-point Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree), with higher scores indicating better social support. The MSPSS has good psychometric properties and used among students (Dambi et al., 2018).
Social support | Three months after training completes
  Social support will be measured using the Multidimensional Scale of Perceived Social Support Scale (MSPSS, Zimet et al., 1988). Items are rated on a 7-point Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree), with higher scores indicating better social support. The MSPSS has good psychometric properties and used among students (Dambi et al., 2018).
Learning | Baseline
  Students' learning will be measured during the Motivated Strategies for Learning Questionnaire (MSLQ, Pintrich et al., 1991). The following subscales from MSLQ will be used: (1) Control of learning beliefs, (2) self-efficacy, (3) test anxiety, (4) meta-cognitive self-regulation, (5) time and study environment and (6) effort regulation. Items are rated on a 7-point Likert scale ranging from 1 (Not true at all of me) to 7 (very true of me), with higher scores indicating better learning strategies.
Learning | After training completes
  Students' learning will be measured during the Motivated Strategies for Learning Questionnaire (MSLQ, Pintrich et al., 1991). The following subscales from MSLQ will be used: (1) Control of learning beliefs, (2) self-efficacy, (3) test anxiety, (4) meta-cognitive self-regulation, (5) time and study environment and (6) effort regulation. Items are rated on a 7-point Likert scale ranging from 1 (Not true at all of me) to 7 (very true of me), with higher scores indicating better learning strategies.
Learning | Three months after training completes
  Students' learning will be measured during the Motivated Strategies for Learning Questionnaire (MSLQ, Pintrich et al., 1991). The following subscales from MSLQ will be used: (1) Control of learning beliefs, (2) self-efficacy, (3) test anxiety, (4) meta-cognitive self-regulation, (5) time and study environment and (6) effort regulation. Items are rated on a 7-point Likert scale ranging from 1 (Not true at all of me) to 7 (very true of me), with higher scores indicating better learning strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lau, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong